CLINICAL TRIAL: NCT01118468
Title: Systematic Assessment of Competitive Flow in Coronary Artery Bypass Grafts by Wave Intensity Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 1426
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Bypass
Keywords: Competitive Flow; Coronary artery bypass; Wave Intensity Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Narrowing of the arteries that supply blood to the heart can lead to heart attacks and death. One way of treating this is to use artery and vein grafts from other parts of the body to bypass the narrowing. However, the blood flow from these grafts "competes" with flow through the natural coronary artery. This may contribute to grafts narrowing with time. This protocol aims to determine the pressure changes responsible for this effect. This could improve our understanding of why some grafts last longer than others.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous coronary artery bypass grafts undergoing coronary angiography and graft restudy

Exclusion Criteria:

* Patient's with cardiac pacemakers, valvular heart disease, and chronic renal failure
* Unable to consent
* Contraindications to adenosine
* Contraindications to cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previous bypass grafts undergoing angiography/ angioplasty who meet stduy criteria
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Davies, MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, United Kingdom